CLINICAL TRIAL: NCT02268812
Title: Patient Registry of Intrathecal Pain Management in Europe: An Open-label, Long-term, Multi-center, Multi-national Post-marketing Observational Study of the Use of Prialt (Ziconotide Intrathecal Infusion) and Alternative Drugs for the Management of Severe, Chronic Pain.
Brief Title: Patient Registry of Intrathecal Pain Management in Europe for Prialt (Ziconotide Intrathecal Infusion) and Alternative Drugs for the Management of Severe, Chronic Pain.
Acronym: PRIME
Status: Completed | Type: Observational
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: SNX-111-E044-401
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-01

CONDITIONS: Pain Management; Severe Chronic Pain
Keywords: Pain Management; Europe; Intrathecal
MeSH Terms: conditions — Agnosia; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ziconotide: No drug will be provided by the sponsor. Treatment decisions will be made by physicians independent of participation in the registry.
  IT analgesia may consist of ziconotide or any other drug used in IT therapy, including those used off-label as part of local clinical practice.

SUMMARY:
This is an open-label, long-term, multi-center multi-national post-marketing observational registry. The objective of this study is to monitor the long-term efficacy, safety, tolerability and quality of life outcomes associated with ziconotide (Prialt) and other analgesics utilized in the intrathecal (IT) management of severe chronic pain.

DETAILED DESCRIPTION:
This is an observational non-interventional registry. All patients will sign and date an Informed Consent Form (ICF) before enrollment (Baseline Visit). Normal clinical practice will be followed. Patients will continue to follow their usual schedule of clinic visits as determined by their physician, during which information and patient-completed questionnaires will be collected (at scheduled intervals timed to coincide with pump refill).

ELIGIBILITY:
Inclusion Criteria

Patients will be eligible to enroll onto the registry if they have given informed consent and meet the following criteria:

* Patient's physician has deemed that the initiation/switch of intrathecal analgesia appropriate, or patient is presently utilizing ziconotide (Prialt)
* Patient has a diagnosis of severe, chronic pain for which intrathecal infusion is indicated
* Patient is at least 18 years of age at time of study entry

All patients starting ziconotide (Prialt) should comply with the indications and warnings in the current approved version of the Summary of Product Characteristics (SmPC).

Exclusion Criteria

Patients who meet any of the following criteria will not be eligible to enroll in the registry:

* Patient is a pregnant or lactating female
* Patient is receiving intrathecal chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have a diagnosis of severe, chronic pain for which intrathecal infusion is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Ziconotide Monotherapy: Participants who took ziconotide alone.
- Ziconotide Combination: Participants who took ziconotide in combination with another intrathecal (IT) therapy.
- Other IT Monotherapy: Participants who took an IT therapy other than ziconotide.
- Other IT Combination: Participants who took two (or more) IT therapies in conjunction other than ziconotide.
Period: Overall Study
Arm/Group | Ziconotide Monotherapy | Ziconotide Combination | Other IT Monotherapy | Other IT Combination
Started | 77 | 72 | 30 | 40
Completed | 61 | 40 | 21 | 26
Not Completed | 16 | 32 | 9 | 14
Not completed — Adverse Event | 8 | 26 | 7 | 10
Not completed — Protocol deviation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Physician Decision | 3 | 1 | 0 | 1
Not completed — Other | 5 | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants who had at least one dose of an intrathecal (IT) therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziconotide Monotherapy | Ziconotide Combination | Other IT Monotherapy | Other IT Combination | Total
Number analyzed (Participants) | 77 | 72 | 30 | 40 | 219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.2 (11.56) | 55.9 (13.46) | 56.7 (12.78) | 54.4 (11.69) | 54.8 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 11 | 18 | 89
  Male | 45 | 44 | 19 | 22 | 130

OUTCOME MEASURES:

1. Primary Outcome: Average Overall Change From Baseline (Visit 1) in Visual Analog Scale of Pain Intensity (VASPI)
Description: VASPI is a worldwide validated measure of pain intensity. A Visual Analog Score (VAS) for pain is determined by using a horizontal line, 100-millimeter (mm) in length, anchored by word descriptors at each end; "no pain" (0 mm) on the left end and "worst imaginable pain" (100 mm) on the right end. The participant was asked to mark on the line the point that they feel represents their current state of pain. A VAS for least pain (over last two weeks), usual pain (over last two weeks), and pain today was determined and averaged to derive the total VAS score ranging from 0 (no pain) to 100 (worst pain imaginable). A last observation carried forward (LOCF) dataset was used to account for missing data where First Visit data could be carried forward.
Time Frame: Month 8 (Visit 4), Month 12 (Visit 5), and Termination Visit (12 months after last participant was enrolled)
Population: Intent-to-Treat (ITT) (LOCF) population included all participants who had at least one dose of an IT therapy. Total number of participants for the outcome measures (335) does not match the total number enrolled (219) due to participants switching between treatment arms as allowed per protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ziconotide Monotherapy | Ziconotide Combination | Other IT Monotherapy | Other IT Combination
Number analyzed (Participants) | 83 | 114 | 67 | 71
Units on a scale
  Month 8 (Visit 4) | -3.23 (23.160) | -15.24 (23.614) | -1.50 (20.736) | -18.40 (21.899)
  Month 12 (Visit 5) | -3.78 (23.424) | -9.33 (30.039) | 1.67 (20.894) | -14.33 (29.800)
  Termination Visit | -6.01 (23.220) | 0.65 (28.208) | 1.64 (21.643) | -14.27 (34.620)

2. Secondary Outcome: Overall Change in Pain Severity and Pain Interference From Baseline (Visit 1) to Month 12 (Visit 5)
Description: The Brief Pain Inventory-Short Form (BPI-SF) survey is made up of two dimensions: pain intensity/severity and pain interference, with each dimension containing specific items that are graded (e.g. mood, walking ability, relations with other people, enjoyment of life, etc.). Each item was graded on an 11-point Likert scale. The pain intensity/severity survey was used to measure pain severity, where 0 was "no pain" and 10 was "pain as bad as you can imagine" for each item listed. The pain interference survey scored each item on a scale, where 0 was "does not interfere" to 10 was "completely interferes". The change in pain severity and pain interference from Baseline (Visit 1) were calculated from the scores.
Time Frame: Baseline (Visit 1) to Month 12 (Visit 5)
Population: ITT LOCF population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziconotide Monotherapy | Ziconotide Combination | Other IT Monotherapy | Other IT Combination
Number analyzed (Participants) | 83 | 114 | 67 | 71
Scores on a scale
  Pain severity | -0.41 (1.768) | -0.77 (2.150) | -0.09 (1.741) | -0.99 (1.866)
  Pain interference | -0.52 (1.645) | -0.42 (2.445) | -0.43 (2.248) | -0.33 (2.039)

3. Secondary Outcome: Overall Change in Pain Severity and Pain Interference From Baseline (Visit 1) to Termination Visit
Description: The BPI-SF survey is made up of two dimensions: pain intensity/severity and pain interference, with each dimension containing specific items that are graded (e.g. mood, walking ability, relations with other people, enjoyment of life, etc.). Each item was graded on an 11-point Likert scale. The pain intensity/severity survey was used to measure pain severity, where 0 was "no pain" and 10 was "pain as bad as you can imagine" for each item listed. The pain interference survey scored each item on a scale, where 0 was "does not interfere" to 10 was "completely interferes". The change in pain severity and pain interference from Baseline (Visit 1) were calculated from the scores.
Time Frame: Baseline (Visit 1) to Termination Visit (12 Months after last participant was enrolled)
Population: ITT LOCF population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziconotide Monotherapy | Ziconotide Combination | Other IT Monotherapy | Other IT Combination
Number analyzed (Participants) | 83 | 114 | 67 | 71
Scores on a scale
  Pain severity | -0.27 (2.219) | -1.11 (2.127) | -0.04 (1.957) | -0.74 (2.321)
  Pain interference | -0.77 (2.809) | -1.05 (2.798) | -0.73 (1.718) | -0.72 (2.054)

4. Secondary Outcome: Number of Participants Who Experienced at Least One Treatment-Emergent Adverse Event (TEAE)
Description: Safety assessments consisted of monitoring and recording all adverse events (AEs) and serious adverse events (SAEs), any therapeutic interventions including all drug therapies, vital signs, and creatine kinase (CK) if laboratory tests were taken by the physician as part of routine clinical practice. AEs were graded on a 3-point scale; 1) mild - discomfort noticed, but no disruption of normal daily activity, 2) moderate - discomfort sufficient to reduce or affect normal daily activity, 3) severe - incapacitating, with inability to work or to perform normal daily activity. A TEAE was defined as an adverse event (AE) with a start date on or after the date of the First Visit. Where a start date was missing, the AE was considered to be treatment-emergent.
Time Frame: From first dose up to 30 days after the last dose of study treatment, for up to approximately 4 years 4 months.
Population: Safety population included all participants who had at least one dose of an IT therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Ziconotide Monotherapy | Ziconotide Combination | Other IT Monotherapy | Other IT Combination
Number analyzed (Participants) | 83 | 114 | 67 | 71
Participants
  Any TEAEs | 66 | 88 | 46 | 48
  Drug-related TEAEs | 56 | 54 | 26 | 28
  SAEs | 26 | 51 | 24 | 30
  Drug-related SAEs | 7 | 11 | 9 | 5
  TEAEs leading to death | 3 | 26 | 7 | 12

5. Other Pre Specified Outcome: Changes in Primary Intrathecal Drug, Including Dose Adjustment and Intervals
Description: Data for this outcome measure was collected as part of the participant's study visit, however was not analyzed as an efficacy endpoint for reporting.
Time Frame: 12 months after the last patient was enrolled
Population: Data for this outcome measure was collected as part of the participant's study visit, however was not analyzed as an efficacy endpoint for reporting.
Arm/Group | Ziconotide Monotherapy | Ziconotide Combination | Other IT Monotherapy | Other IT Combination
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Other Pre Specified Outcome: Change in the Actual Overall EuroQoL (EQ-5D) Health Score From First Visit to Month 12 and End of Study
Description: The EQ-5D is a standardized instrument used to measure quality of life. It classifies health states across five domains: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each domain has three levels (no problems, some/moderate problems, extreme problems). A unique EQ-5D health state was defined by combining one level from each of the five dimensions. The response to the question of how good or bad the participant's health was today was given on a visual analogue scale of 0 to 100 millimeters (mm), where 0 meant the participant was in the worst imaginable health state today and 100 meant the participant was in the best imaginable health state today. The results for the Health Score were that of the calculated overall score of the five dimensions, where -0.594 is worst health and 1.00 is perfect health. Change is defined as change in actual from the First Visit.
Time Frame: Month 12 Visit, End of Study (Termination Visit)
Population: ITT population. Missing items/values used in calculating the partially complete Health Score were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziconotide Monotherapy | Ziconotide Combination | Other IT Monotherapy | Other IT Combination
Number analyzed (Participants) | 83 | 114 | 67 | 71
Scores on a scale
  Month 12: number analyzed (Participants) | 21 | 12 | 15 | 8
  Month 12 | -0.01 (0.176) | -0.06 (0.207) | 0.01 (0.217) | -0.01 (0.136)
  End of Study: number analyzed (Participants) | 33 | 15 | 22 | 22
  End of Study | -0.00 (0.196) | 0.04 (0.180) | -0.03 (0.193) | -0.02 (0.145)

ADVERSE EVENTS:
Time Frame: For each participant, from the first dose till 30 days after the last dose or up to the termination visit (which was 12 months after the last subject had been enrolled), or approximately 4 years.
Description: The safety population included all participants who received at least one dose of an IT therapy. Treatment emergent adverse events (TEAEs) and serious adverse events were reported. Participants could switch IT therapies during the study, so AEs were assigned to the treatment taken at the time and date of the onset of the AE. This resulted in the possibility of a participant being counted in more than one therapy category.
Arm/Group | Ziconotide Monotherapy | Ziconotide Combination | Other IT Monotherapy | Other IT Combination
All-Cause Mortality (participants affected / at risk) | 3/83 | 26/114 | 7/67 | 12/71
Serious Adverse Events (participants affected / at risk) | 26/83 | 51/114 | 24/67 | 30/71
Other Adverse Events (participants affected / at risk) | 59/83 | 70/114 | 34/67 | 43/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziconotide Monotherapy (N=83) | Ziconotide Combination (N=114) | Other IT Monotherapy (N=67) | Other IT Combination (N=71)
Death (General disorders) | 0 | 7 | 7 | 2
Pain (General disorders) | 0 | 4 | 3 | 3
General Physical Health Deterioration (General disorders) | 0 | 4 | 1 | 2
Catheter Related Complication (General disorders) | 0 | 1 | 0 | 3
Pyrexia (General disorders) | 1 | 2 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1 | 1 | 0
Catheter Site Pain (General disorders) | 0 | 0 | 1 | 0
Disease Progression (General disorders) | 1 | 0 | 0 | 0
Drug Withdrawal Syndrome (General disorders) | 0 | 0 | 0 | 1
Extravasation (General disorders) | 0 | 1 | 0 | 0
Face Oedema (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Generalised Oedema (General disorders) | 0 | 1 | 0 | 0
Infusion Site Mass (General disorders) | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 4 | 2 | 4
Meningitis (Infections and infestations) | 1 | 0 | 2 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 2 | 0
Catheter Related Infection (Infections and infestations) | 0 | 0 | 1 | 2
Device Related Infection (Infections and infestations) | 2 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Breast Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Implant Site Infection (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Rectal Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Soft Tissue Infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal Skin Infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Non-small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Bone Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colorectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Medical Device Complication (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Device Dislocation (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Device Connection Issue (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Inadequate Analgesia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Suture Related Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound Secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 3 | 0 | 0
Depression (Psychiatric disorders) | 0 | 4 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 1 | 1 | 0
Mental Disorder (Psychiatric disorders) | 1 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Drug Abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucinations, Mixed (Psychiatric disorders) | 0 | 1 | 0 | 0
Hostility (Psychiatric disorders) | 0 | 0 | 1 | 0
Narcissistic Personality Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Head Titubation (Nervous system disorders) | 0 | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Speech Disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1 | 0 | 0
Stupor (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Trigeminal Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Shock Haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 1
Circulatory Collapse (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Venous Occlusion (Vascular disorders) | 0 | 0 | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchial Secretion Retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 1 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Feeding Disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 3 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Central Venous Catheterisation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Drug Therapy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Medical Device Removal (Surgical and medical procedures) | 1 | 0 | 0 | 0
Nerve Block (Surgical and medical procedures) | 0 | 1 | 0 | 0
Peripheral Nerve Decompression (Surgical and medical procedures) | 1 | 0 | 0 | 0
Spinal Nerve Stimulator Implantation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 1
C-reactive Protein Increased (Investigations) | 0 | 1 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Behcet's Syndrome (Immune system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Biliary Dilatation (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Skin Erosion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziconotide Monotherapy (N=83) | Ziconotide Combination (N=114) | Other IT Monotherapy (N=67) | Other IT Combination (N=71)
Dizziness (Nervous system disorders) | 15 | 6 | 5 | 3
Headache (Nervous system disorders) | 11 | 5 | 5 | 8
Memory Impairment (Nervous system disorders) | 10 | 8 | 0 | 0
Somnolence (Nervous system disorders) | 3 | 4 | 3 | 4
Hypoaesthesia (Nervous system disorders) | 4 | 0 | 1 | 7
Nausea (Gastrointestinal disorders) | 15 | 5 | 10 | 10
Constipation (Gastrointestinal disorders) | 6 | 7 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 3 | 2
Dry Mouth (Gastrointestinal disorders) | 5 | 4 | 2 | 3
Vomiting (Gastrointestinal disorders) | 2 | 3 | 3 | 4
Oedema Peripheral (General disorders) | 5 | 5 | 4 | 6
Fatigue (General disorders) | 6 | 3 | 6 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 3 | 2 | 8
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 5 | 4 | 2 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 4 | 2 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 6
Confusional State (Psychiatric disorders) | 5 | 6 | 2 | 1
Insomnia (Psychiatric disorders) | 6 | 1 | 1 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 5 | 9 | 7
Weight Decreased (Investigations) | 5 | 1 | 3 | 4
Vertigo (Ear and labyrinth disorders) | 3 | 6 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less